CLINICAL TRIAL: NCT05996016
Title: A Cohort Study Among HIV Infected Women：Exploring the Regulatory Mechanism of Gut and Vaginal Microbiota in HPV Infection and Cervical Lesion
Brief Title: Gut and Vaginal Microbiota Profile Study for HIV Women
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PekingUMCH-K2675
Record Dates: First submitted 2022-11-28; First posted 2023-08-16 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-10

CONDITIONS: HPV; HIV Infections; Vaginal Microbiota
Keywords: HPV; Women With HPV infection; vaginal microbiota; gut microbiota
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
Women Living with HIV Infection （WLHIV）are intended to acquire HPV infection which usually contributes to variable cervical lesions. we hypothesize that vaginal microbiota imbalance may make WLHIV prone to HPV infection，thereafter results in severe cervical lesion.

DETAILED DESCRIPTION:
Women Living with HIV Infection （WLHIV）are intended to acquire HPV infection which usually contributes to variable cervical lesions. Besides the HPV co-infection, microbiota study recently reveals that the changes of vaginal bacteria spectrum might also be related with cervical disease in WLHIV. However, data on HPV prevalence in WLHIV and its associated cervical lesion incidence is still limited in China. Moreover, the causal relationship between vaginal microbiota and cervical lesion in WLHIV is not clear. Here, we hypothesize that vaginal microbiota imbalance may make WLHIV prone to HPV infection，thereafter results in severe cervical lesion.

ELIGIBILITY:
Inclusion Criteria:

* HIV women （including pregnant）;
* sign consent paper

Exclusion Criteria:

* virgin or maiden

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women with HIV Infection from 6 HIV care centers across CHINA, including Beijing, Zhejiang, Guangxi, Yunan, Shanxi and Shandong.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
HPV infection incidence | 0, 6m, 12m, 24m, 36m
  To collect 400 analyzable samples from women with HIV, including HPV screening, fecal and vaginal microflora samples. Cervical HPV screening will be collected as required in standard containers and stored for transport to the central laboratory.the rates of HPV infection.
cervical lesions | 0, 6m, 12m, 24m, 36m
  To collect 400 analyzable samples from women with HIV, including vaginal cleanliness assessment and TCT examination. vaginal swab samples will be collected as required in standard containers and stored for transport to the central laboratory.Variable cervical lesions, including CIN I-III and neoplasma.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Lyu, MD, Principal Investigator — No. 10Yi，Chaowai Street ，Chaoyang District ，Beijing ，China
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No